CLINICAL TRIAL: NCT00736268
Title: Telephone-based Intervention for Patients With COPD and Their Caregivers
Brief Title: Coping Skills for Patients With Chronic Obstructive Pulmonary Disease (COPD) and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00003707; 2R01HL065503-06A1 (NIH)
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung Disease; Chronic Bronchitis; Emphysema; Caregiver stress; COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Bronchitis, Chronic; Emphysema; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CST (Experimental): Telephone-based Enhanced Coping Skills Training (CST)
  Interventions: Behavioral: Telephone-based Enhanced Coping Skills Training (CST)
- UMC (Other): Usual Medical Care and COPD education and symptom monitoring (UMC)
  Interventions: Other: Usual Medical Care and COPD education and symptom monitoring (UMC)

INTERVENTIONS:
Behavioral: Telephone-based Enhanced Coping Skills Training (CST) — Telephone-based Enhanced Coping Skills Training (CST) intervention will systematically train participants (and caregivers) in the use of coping skills for symptom management (i.e. activity pacing, pleasant activity scheduling, communications, relaxation, goal setting, imagery, calming self-statements, problem solving, and preventing and dealing with setbacks). Participants in the CST condition will receive 12 weekly 30 minute telephone sessions followed by 2 bi-weekly booster sessions for training in symptom management strategies. Participants and caregivers will be evaluated at baseline, at the conclusion of 4 months of treatment, and at annual follow-up intervals for up to 4 years.
  Arms: CST
Other: Usual Medical Care and COPD education and symptom monitoring (UMC) — COPD usual care plus education and symptom monitoring control condition will participate in a weekly 15 minute phone call followed by 2 bi-weekly phone calls, assessing their health status and providing them with support and COPD education. COPD Education topics include types of lung disease, oxygen use, medication management, preventing infection, managing daily activities, and nutrition. Participants and caregivers will be evaluated at baseline, at the conclusion of 4 months of treatment, and at annual follow-up intervals for up to 4 years.
  Arms: UMC

SUMMARY:
This study is an NIH-funded clinical trial conducted at Duke University Medical Center and Ohio State University. The purpose of this study is to examine the effects of a telephone-based, care-giver assisted, coping skills training (CST) program in patients with Chronic Obstructive Pulmonary Disease (COPD) and their caregivers. This may help COPD patients and their caregivers to deal better with the stress of lung disease. This study will test 3 primary hypotheses: 1) That enhanced CST will be more effective in improving quality of life compared to a Usual Medical Care plus COPD education and symptom management control group; 2) That enhanced CST will be associated with better medical outcomes (i.e., greater survival and fewer COPD-related physician visits or hospitalizations) compared to Controls over a follow-up period of up to 4 years; and 3) That improvements in quality of life and survival will be mediated by increased functional capacity and better coping.

This proposed study builds upon our prior research by: a) adapting and refining our CST protocol, which was effective in improving psychosocial adjustment in patients awaiting lung transplantation, to a broader population of patients with COPD who are not immediate candidates for lung transplantation; b) enhancing our intervention to improve functional capacity, reduce somatic symptoms, and improve survival; c) examining the impact of CST on medical expenditures; and d) including caregivers in an enhanced CST intervention.

DETAILED DESCRIPTION:
Overall, 746 participants (patients and caregivers) were consented for participation into this study from both Duke University Medical Center and Ohio State University. Of these, 326 patients were randomized and participated in the study intervention along with 252 consented participants who acted as a caregiver; in total 578 participants (patients and caregivers) were involved with the study intervention.

ELIGIBILITY:
Inclusion Criteria:

* male or female outpatients 21 years of age or older
* a diagnosis of COPD
* FEV1 25%-80% of predicted value
* FEV1/FVC <70%
* capacity to give informed consent and follow study procedures

Exclusion Criteria:

* dementia
* psychotic features including delusions or hallucinations
* acute suicide or homicide risk
* other illness (e.g., cancer) that is likely to cause death within 3 years
* unstable angina
* congestive heart failure stage III - IV by NYHA classification
* active involvement in pulmonary rehabilitation or a formal exercise program

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2008-08; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Composite measure of psychological quality of life, composite index of all cause mortality and COPD-related hospitalization. | 4 years

SECONDARY OUTCOMES:
Composite measure of somatic quality of life | 4 months and up to 4 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Blumenthal JA, Babyak MA, Keefe FJ, Davis RD, Lacaille RA, Carney RM, Freedland KE, Trulock E, Palmer SM. Telephone-based coping skills training for patients awaiting lung transplantation. J Consult Clin Psychol. 2006 Jun;74(3):535-44. doi: 10.1037/0022-006X.74.3.535. PMID 16822110
- [Background] Martinu T, Babyak MA, O'Connell CF, Carney RM, Trulock EP, Davis RD, Blumenthal JA, Palmer SM; INSPIRE Investigators. Baseline 6-min walk distance predicts survival in lung transplant candidates. Am J Transplant. 2008 Jul;8(7):1498-505. doi: 10.1111/j.1600-6143.2008.02264.x. PMID 18510641
- [Background] Emery CF, Leatherman NE, Burker EJ, MacIntyre NR. Psychological outcomes of a pulmonary rehabilitation program. Chest. 1991 Sep;100(3):613-7. doi: 10.1378/chest.100.3.613. PMID 1889242
- [Derived] Blumenthal JA, Emery CF, Smith PJ, Keefe FJ, Welty-Wolf K, Mabe S, Martinu T, Johnson JJ, Babyak MA, O'Hayer VF, Diaz PT, Durheim M, Baucom D, Palmer SM. The effects of a telehealth coping skills intervention on outcomes in chronic obstructive pulmonary disease: primary results from the INSPIRE-II study. Psychosom Med. 2014 Oct;76(8):581-92. doi: 10.1097/PSY.0000000000000101. PMID 25251888